CLINICAL TRIAL: NCT01938014
Title: Lysosomal Storage Disease: Health, Development, and Functional Outcome Surveillance in Preschool Children
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other); State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Other Study IDs: RDCRN-LDN-6710; U54NS065768 (NIH)
Record Dates: First submitted 2013-08-06; First posted 2013-09-10 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Mucopolysaccharidosis Type I (MPS I); Mucopolysaccharidosis Type II (MPS II); Mucopolysaccharidosis Type III (MPS III); Mucopolysaccharidosis Type VI (MPS VI); Krabbe Disease
Keywords: MPS I; MPS II; MPS III; MPS VI; Krabbe disease; globoid cell leukodystrophy; galactosylceramide lipidosis; mucopolysaccharidoses; mucopolysaccharidosis; Rare Diseases Clinical Research Network; Lysosomal Disease Network; enzyme replacement therapy; hematopoietic stem cell transplant; telephone-based surveillance; Hurler syndrome; Hunter syndrome; Scheie syndrome; Hurler-Scheie syndrome; Sanfilippo syndrome; Maroteaux-Lamy syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Sudden Infant Death; Mucopolysaccharidosis III; Mucopolysaccharidosis VI; Leukodystrophy, Globoid Cell; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None collected; this is data-collection only, via a telephone-interview of children's care-givers.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothesis: Children diagnosed with a lysosomal disease will exhibit developmental, adaptive, and behavioral strengths and difficulties depending upon 1) biomedical risk factors (i.e. the specific genetic disorder responsible for the illness); 2) available modifying interventions, whether medical or behavioral; and 3) social risks in the children's families, neighborhoods and communities. A valid and reliable telephone-based surveillance system can successfully collect the data required to elucidate these developmental, adaptive and behavioral strengths and difficulties.

DETAILED DESCRIPTION:
Children who have lysosomal disease experience declines in health status and central nervous system integrity which result in motor, communication, self-care, learning and behavioral challenges. Medical interventions such as enzyme replacement therapy (ERT) and hematopoietic stem cell transplantation can improve the health and functioning of children with lysosomal disease. To date, however, there is no established system for evaluating the health status, developmental status, behavioral outcomes or functional outcomes of these preschool-aged children across time and differing settings. The primary objective of this study is to develop a valid and reliable telephone-based data-gathering system for obtaining health status data, developmental status data, behavioral outcomes data, and functional outcomes data which reflect skills of daily living including feeding, moving, communicating and responding to others.

The secondary objective of this study is to assess the validity of several early-childhood standardized assessment tools as compared to the standard neuropsychological assessment battery specified by the Lysosomal Disease Network's 'Neurobehavioral Core.'

The third objective of this study is to describe the impact of lysosomal disease upon the families of lysosomal disease-affected children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 1 to 84 months who have been diagnosed with MPS types I, II, III or VI. Children aged 1 to 84 months who have been diagnosed with some other lysosomal disease. Children aged birth to 18 years who have been diagnosed with Krabbe disease, or who have a positive screening for Krabbe disease.

Exclusion Criteria:

Children who do not have a lysosomal disease are excluded from this study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Children aged 1 to 84 months who have been diagnosed with MPS types I, II, III or VI
  2. Children aged 1 to 84 months who have been diagnosed with some other lysosomal disease
  3. Children aged birth to 18 years who have been diagnosed with Krabbe disease, or who have a positive screening for Krabbe disease
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2016-07-23 (Actual); Study Completion 2016-07-23 (Actual)

PRIMARY OUTCOMES:
Change in Health Status of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the lysosomal disease-affected child's health status.

SECONDARY OUTCOMES:
Change in the Behavioral Outcomes of the Immediate Family of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the behavioral outcomes of the immediate family of the lysosomal disease-affected child.
Change in Developmental Status of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the lysosomal disease-affected child's developmental status.
Change in Behavioral Outcomes of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the lysosomal disease-affected child's behavioral outcomes.
Change in Functional Outcomes of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the lysosomal disease-affected child's functional outcomes.
Change in the Functional Outcomes of the Immediate Family of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the functional outcomes of the immediate family of the lysosomal disease-affected child.
Change in the Well-Being of the Immediate Family of the Lysosomal Disease-Affected Child Measured at 6-month Intervals for 5.5 Years | Upon Enrollment, and thereafter at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 months post-enrollment
  Using the technique of telephone-based interviews with the child's care-giver(s), the investigators will obtain and record verbal responses to a variety of standardized assessment tools which seek to ascertain the state of well-being of the immediate family of the lysosomal disease-affected child.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Msall, M.D., Principal Investigator — University of Chicago; Patricia K. Duffner, M.D., Principal Investigator — Hunter James Kelly Institute in Buffalo, New York; Chester B. Whitley, Ph.D., M.D., Principal Investigator — University of Minnesota; Nancy Lyon, CPNP, Principal Investigator — Hunter James Kelly Institute in Buffalo, New York
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Hunter James Kelly Institute, Buffalo, New York

REFERENCES:
- See also: Rare Diseases Clinical Research Network — https://www.rarediseasesnetwork.org
- See also: Hunter James Kelly Research Institute — http://hjkri.buffalo.edu/